CLINICAL TRIAL: NCT02836561
Title: Contraceptive Choice at the Time of Uterine Evacuation: A Randomized Controlled Pre-visit LARC Educational Intervention
Brief Title: Contraceptive Choice at the Time of Uterine Evacuation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Planned Parenthood League of Massachusetts (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2016P000619
Record Dates: First submitted 2016-06-17; First posted 2016-07-19 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Contraception

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Message (Experimental): Participants who are randomized to the intervention message will receive contraception information in advance of their appointment that may be helpful in their decision-making.
  Interventions: Other: Telephone message
- Control Message (No Intervention): Participants who are randomized to the control message will receive appointment logistic information that may be a helpful reminder.

INTERVENTIONS:
Other: Telephone message — A pre-visit telephone intervention describing availability of long-acting reversible contraceptives at time of uterine evacuation
  Arms: Intervention Message

SUMMARY:
The goal of this project is to investigate whether a pre-visit telephone intervention could increase awareness of long-acting reversible contraception (LARC) availability at the time of uterine evacuation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Scheduled for uterine evacuation
* Speaks English proficiently in order to understand the telephone conversation and the survey questions.

Exclusion Criteria:

* Previous participation in this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2016-07; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Knowledge that LARC can start at uterine evacuation: Percentage of women who report that LARC methods are available to start at the time of uterine evacuation, as assessed on a questionnaire created for this study | Day 1: Questionnaire administered prior to the information session
  Percentage of women who know that the implant and IUD are available to start at the time of uterine evacuation, as assessed on a questionnaire created for this study. Compared between those who receive the pre-visit information (intervention group) and those who do not receive this information (control group)

SECONDARY OUTCOMES:
Intervention utility: Percentage of women who report that receiving information about contraception before their appointment was either very useful or somewhat useful, as assessed on a 4-point scale on a questionnaire created for this study | Day 1: Questionnaire administered prior to information session
  Percentage of women who who report that receiving information about contraception before their appointment was either very useful or somewhat useful, as assessed on a 4-point scale on a questionnaire created for this study. Compared between those who received pre-visit information about contraception (intervention group) and those who did not (control group)
General LARC knowledge: Percentage of women with a high score (cutpoint to be determined) on a 10-question LARC knowledge scale developed for this study | Day 1: Questionnaire administered prior to information session
  Percentage of women with a high score (cutpoint to be determined) on a 10-question LARC knowledge scale developed for this study. Compared between those who received the pre-visit information about contraception (intervention group) and those who did not (control group)
Intent to use LARC: Percentage of women who report a LARC method as their preferred method of birth control, as assessed on a questionnaire created for this study | Day 1: Questionnaire administered prior to information session
  Percentage of women who report a LARC method as their preferred method of birth control, as assessed on a questionnaire created for this study. Compared between those who received the pre-visit information about contraception (intervention group) and those who did not (control group)
LARC stage of change: Percentage of women who report being somewhat or very interested in starting a LARC method, as assessed on a 4-point scale on a questionnaire created for this study | Day 1: Questionnaire administered prior to information session
  Percentage of women who report being somewhat or very interested in starting an implant or IUD, as assessed on a 4-point scale on a questionnaire created for this study. Compared between those who received pre-visit information about contraception (intervention group) and those who did not (control group)
Uptake of LARC at time of uterine evacuation: Percentage of women who receive a LARC method at the time of uterine evacuation, as documented within the electronic medical record | Day 1: Data abstraction to be performed after the subject's day 1 visit complete
  Percentage of women who receive an implant or an IUD at the time of uterine evacuation, compared between those who received pre-visit information about contraception (intervention group) and those who did not (control group)

CONTACTS AND LOCATIONS:
Overall Officials: Principal Investigator, MD, Principal Investigator — Planned Parenthood League of Massachusetts
Locations (1):
- Planned Parenthood League of Massachusetts, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Present at conferences and publish results in peer reviewed journal

REFERENCES:
- [Derived] Roe AH, Fortin J, Gelfand D, Janiak E, Maurer R, Goldberg A. Advance notice of contraceptive availability at surgical abortion: a pilot randomised controlled trial. BMJ Sex Reprod Health. 2018 Jul;44(3):187-192. doi: 10.1136/bmjsrh-2017-200023. Epub 2018 May 18. PMID 30012721